CLINICAL TRIAL: NCT06237192
Title: Multicenter Prospective Study of Safety and Efficacy MRD-associated Non-intensive But Non-interruptive Treatment of Ph-negative Acute Lymphoblastic Leukemia Adult Patients
Brief Title: MRD-associated Non-intensive But Non-interruptive Treatment of Ph-negative Acute Lymphoblastic Leukemia Adult Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RALL-2016m
Record Dates: First submitted 2024-01-03; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRD-positive with Target therapy (Experimental): MRD-positive patients after induction therapy in target therapy group (for B-ALL- blinatumomab, for T-ALL - venetoclax+ChT)
  Interventions: Drug: blinatumomab for B-ALL, venetoclax for T-ALL

INTERVENTIONS:
Drug: blinatumomab for B-ALL, venetoclax for T-ALL — MRD-associated based therapy for Ph-negative acute lymphoblastic leukemia

SUMMARY:
Non-intensive But Non-interruptive Treatment based on previously study RALL-2016 of Adult Ph-negative Acute Lymphoblastic Leukemia: No high-dose methotrexate (MTX) and high-dose cytarabine (ARA-C) consolidation blocks, L-asparaginaseis scheduled for 1 year of treatment, 21 intrathecal injections through the whole treament, T-ALL patients in complete remission (CR) with MRD-positive status after 2nd induction receive consolidation 1-3 with venetoclax (56 days), and B-ALL patients in complete remission (CR) with MRD-positive status after 2nd induction receive 1 consolidation with blinatumomab. After that consolidation bone samples are collected and tested for MRD and patients will continue therapy by protocol without HSCT if MRD-negative (by flow cytometry by aberrant immunophenotype in a centralized lab) status was achieved.

DETAILED DESCRIPTION:
* 7 days prednisolone prephase
* 8 weeks induction with de-escalation of induction chemotherapy: 3 instead of 4 dauno/vncr pulses,

  1. instead of 2 Cph injections during induction,
  2. instead of 4 ARA-C blocks, distribution of of L-asp injections through all phases
* After CR achievement T-cell ALL and B-ALL patients are being study MRD (by FCM) MRD-positive patients with T-ALL will receive 1-3 consolidation with venetoclax (400 mg/d), and B-ALL patients will receive1 additional consolidation by blinatumomab
* Non-interruptive 5 consolidation phases with dose modification according to WBC and platelets count after CR achievement. Rotation of consolidation is permitted
* 2 years maintenance for all patients
* 21 TIT through the whole treatment with higher intensity during induction|consolidation
* Centralized MRD monitoring at +70 d, + 133 d, + 190 days; before and after allo-HSCT
* Allo-HSCT is planned only for very high risk patients (11q23 ALL, MRD positivity after target therapy, ETP T-ALL)

ELIGIBILITY:
Inclusion Criteria:

• age 18-55 years old of patient,

- Clinical diagnosis of non-treated Ph-negative ALL

Exclusion Criteria:

• age more than 55 years old,

* Clinical diagnosis of Ph-positive ALL
* Clinical diagnosis of relapsed/refractory ALL,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3-year
  Rate of Diseases-free survival in MRD-positive ALL patients

SECONDARY OUTCOMES:
MRD-negativity after target therapy | 1 month
  Rate of Minimal Residual Disease negativity after target therapy
Overall survival | 3-yaers OS
  Rate of overall survival in protocol

CONTACTS AND LOCATIONS:
Overall Officials: Elena Parovichnikova, MD, PhD, Study Director — National Research Medical Center for Hematology
Locations (1):
- Olga Aleshina, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No